CLINICAL TRIAL: NCT02058303
Title: Exparel (Bupivacaine Liposome Injectable Suspension) for Distal Upper Extremity Blocks in Orthopedic Surgery
Brief Title: Study of A Long Lasting Local Anesthestic for Hand, Wrist or Finger Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI leaving instutition
Sponsor: Jose Soberon, MD (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Jose Soberon, MD, Anesthesiologist, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04262013
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Hand Injuries; Wrist Injuries; Finger Injuries
Keywords: hand surgery; wrist surgery; finger surgery; anesthesia; regional anesthesia; postoperative pain
MeSH Terms: conditions — Hand Injuries; Wrist Injuries; Finger Injuries; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exparel forearm block (Experimental): Under ultrasound guidance, 3-5 milliliters (mL) Exparel will be injected around the 3 nerves of the forearm prior to surgery. 20-30 mL Mepivacaine will be used for the supraclavicular block following the forearm block.
  Interventions: Drug: Exparel Forearm block
- Bupivacaine supraclavicular block (Active Comparator): Under ultrasound guidance, 20-30 mL 0.5% Bupivacaine will be used for the supraclavicular block.
  Interventions: Drug: Bupivacaine supraclavicular block

INTERVENTIONS:
Drug: Exparel Forearm block — 20-30 mL Mepivacaine will be used for the supraclavicular block following the forearm block.
  Other Names: bupivacaine liposome injectable suspension
  Arms: Exparel forearm block
Drug: Bupivacaine supraclavicular block — 20-30mL 0.5% bupivacaine
  Arms: Bupivacaine supraclavicular block

SUMMARY:
The purpose of this study is to compare Exparel, a new, long-lasting numbing medication and a shorter-acting nerve block to a traditional single-shot nerve block in patients having hand, wrist or finger surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years or older having hand, wrist, or finger surgery
* ability to understand and provide informed consent
* American Society of Anesthesiologists status I-III
* presence of a responsible adult caregiver for 48-72 hours after surgery

Exclusion Criteria:

* patient refusal or inability to provide informed consent
* true allergy, not sensitivity to local anesthetics, midazolam, fentanyl, hydromorphone, propofol
* pregnancy
* hepatic or renal failure
* evidence of infection at or near the proposed needle insertion site
* any sensorimotor deficit of the upper extremity
* BMI greater than or equal to 35
* uncontrolled or severe pulmonary disease
* anticoagulant use (not aspirin or non-steroidal anti-inflammatories)
* chronic pain patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Soberon, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Exparel Forearm Block: Under ultrasound guidance, 3-5 mL Exparel will be injected around the 3 nerves of the forearm prior to surgery. 20-30 mL Mepivacaine will be used for the supraclavicular block following the forearm block.
  Exparel Forearm block: 20-30 mL Mepivacaine will be used for the supraclavicular block following the forearm block.
Period: Overall Study
Arm/Group | Exparel Forearm Block | Bupivacaine Supraclavicular Block
Started | 16 | 21
Completed | 16 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel Forearm Block | Bupivacaine Supraclavicular Block | Total
Number analyzed (Participants) | 16 | 21 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (0) | 62.5 (0) | 62.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Onset of Sensorimotor Block
Description: A blinded study staff member will evaluate the subject after the block is performed. Subjects will be asked to move their hand and will be asked if they can feel a sharp sensation on specific areas of their hand. Once no movement and no feeling is detected, the block is considered successful and the time will be noted.
Time Frame: 30 minutes
Population: Discrepancies are due to a subset of subjects not achieving full blockade at 30 minutes.
Measure: Number; unit: proportion of subjects
Groups:
- Bupivacaine Supraclavicular Block: Under ultrasound guidance, 20-30 milliliters (mL) 0.5% Bupivacaine will be used for the supraclavicular block.
  Bupivacaine supraclavicular block: 20-30mL 0.5% bupivacaine
Arm/Group | Exparel Forearm Block | Bupivacaine Supraclavicular Block
Number analyzed (Participants) | 16 | 21
proportion of subjects
  Median nerve block after 30 minutes | 1.0 | .81
  Ulnar nerve block after 30 minutes | .933 | .818
  Radial nerve block after 30 minutes | 1.0 | .864
  Musculocutaneous nerve block after 30 minutes | .933 | .79

ADVERSE EVENTS:
Arm/Group | Exparel Forearm Block | Bupivacaine Supraclavicular Block
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/21
Other Adverse Events (participants affected / at risk) | 0/16 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes